CLINICAL TRIAL: NCT05504382
Title: Effect of Electroacupuncture Versus Phonophoresis on Refractory Pain in Juvenile Rheumatoid Arthritis
Brief Title: Effect of Electroacupuncture on Refractory Pain in Juvenile Rheumatoid Arthritis: Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohamed Abdelmoneim El Meligy (Other)
Responsible Party: Sponsor-Investigator, Mohamed Abdelmoneim El Meligy, DR. Mohamed Abdelmoeim Ahmed Abo-El-Ros, Egyptian Chinese University
Organization: Egyptian Chinese University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003788
Record Dates: First submitted 2022-08-13; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Juvenile Rheumatoid Arthritis
Keywords: Refractory Pain Juvenile Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant
Masking Description: children suffering from juvenile idiopathic arthritis/oligoarthritic (mainly the knee joint) will participate in the study.
  All children will be randomly assigned into 2 groups of equal numbers A, B using sealed envelopes, 21 children for each group.
  * Study group A: will receive especially electrical acupuncture on the knee joint
  * Study group B: will receive naproxen phonophoresis on the knee joint
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group 1 (Experimental): receive especially electrical acupuncture on the knee joint
  Interventions: Device: naproxen phonophoresis
- study group 2 (Experimental): receive naproxen phonophoresis on the knee joint
  Interventions: Device: naproxen phonophoresis

INTERVENTIONS:
Device: naproxen phonophoresis — transmission of naproxen molecule by therapeutic ultrasound
  Other Names: electroacupuncture

SUMMARY:
the purpose of the study is to investigate the effect of Electrical Acupuncture Versus naproxen phonophoresis on Refractory pain in Juvenile Rheumatoid arthritis

DETAILED DESCRIPTION:
Juvenile idiopathic arthritis (JIA) is the most common chronic rheumatic disease in children and adolescents, affecting approximately one in 1000 children in North America. It is diagnosed in children younger than 16 years of age with arthritis in one or more joints for at least six weeks after other causes have been excluded. Arthritis in JIA is characterized by stiffness, pain and swelling of affected joints. The disease course of JIA may involve flares of increased disease activity or chronic persistent joint inflammation, even into adulthood. Various complications may arise secondary to ongoing disease activity or treatment, including joint damage and deformity, growth abnormalities and osteoporosis with fragility fractures The prevalence of refractory pain in children with arthritis is of particular concern because it often contributes to poor physical and psychosocial outcomes. Increased daily symptoms of pain predict considerable functional disability, including significantly reduced participation in school, social and physical activities, and augmented mood disturbance

ELIGIBILITY:
Inclusion Criteria:

* • Age ranges from 14 to 16 years.

  * All children will be assigned to the study are suffering from persistent oligoarthritis.
  * All children have regional knee pain complaint more than 6 weeks.
  * Pain and stiffness especially in the morning, and a joint that feels warm to the touch
  * Low grade fever at the onset of disease

Exclusion Criteria:

* • Neurological disorders.

  * Dermatological disorders.
  * Acute trauma prior to the study.
  * Other co- morbidities like diabetes and conditions associated with inflammation such as malegnancies.
  * Analgesic drugs or NSAIDs during the treatment period.

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
knee pain | 2 weeks
  change in refractory knee pain will be assessed by visual analogue scale

SECONDARY OUTCOMES:
knee joint range of motion | 2 weeks
  change in the range of motion of knee joint will be measured by universal goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abo-El-Ros, Ph.d, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No